CLINICAL TRIAL: NCT01309477
Title: The Efficacy and Tolerance of Tacrolimus Sustained-release Capsules on Refractory Nephrotic Syndrome (RNS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Xueqing Yu, Sun Yat-sen University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSU-PRGNS-002
Record Dates: First submitted 2011-02-01; First posted 2011-03-07 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-10

CONDITIONS: Nephrotic Syndrome
Keywords: Refractory Nephrotic Syndrome; Tacrolimus
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ADVAGRAF (Experimental): All subjects in the study will take the Tacrolimus Sustained-release Capsules (ADVAGRAF) orally at the basis of low dose prednisone treatment
  Interventions: Drug: Tacrolimus Sustained-release Capsules (ADVAGRAF)

INTERVENTIONS:
Drug: Tacrolimus Sustained-release Capsules (ADVAGRAF) — Started: 0.05-0.1mg/kg/d, one time per day, then adjusting the dose to maintain the blood level 5-10ng/ml in the induction treatment .
  Other Names: ADVAGRAF

SUMMARY:
It is a pilot study to explore the efficacy and safety of Tacrolimus Sustained-release Capsules (ADVAGRAF) on 6-month induction therapy of Refractory Nephrotic Syndrome (RNS).

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either sex, 14-60 years of age
* Diagnosis of Nephrotic syndrome with hypoalbuminemia (< 3.0g/dl) and heavy proteinuria (> 3.5g/24hr) and exclude secondary Nephrotic syndrome
* Refractory Nephrotic Syndrome

  1. Steroid resistant: failure to respond (either complete or partial remission) after a course of 8 weeks of 1.0 mg/kg/d prednisone or equal dose of steroid therapy
  2. Steroid dependent: recurrence of nephrotic proteinuria during tapering of prednisone at a dose > 10 mg/day or within the first 2 weeks after withdrawal of prednisone
  3. Frequently recurrence: initial remission with steroid induction therapy, but relapsed 2 or more in 6 months or 3 or more within 12 months
  4. Failure to respond (either complete or partial remission) even after CTX, MMF or CsA therapy combined with steroid
* eGFR ≥ 60 ml/min/1.73 m2
* Provision of written informed consent by subject or guardian

Exclusion Criteria:

* Systemic disease
* eGFR < 60ml/min/1.73m2
* Diagnosed DM
* Malignant tumors (except fully cured basal cell carcinoma)
* Familial nephritic syndrome
* History of significant gastrointestinal disorders (e.g. severe chronic diarrhea or active peptic ulcer disease) within 3 month prior to enter this study
* Any Active systemic infection or history of serious infection within one month of entry or known infection with HIV, hepatitis B, or hepatitis C
* Known hypersensitivity or contraindication to tacrolimus, corticosteroids
* Participation in another clinic trial and/or receipt of investigational drugs within 4 weeks prior to screening
* Pregnancy, nursing or use of a non-reliable method of contraception
* Inability or unwillingness to provide written informed consent
* Usage of immunosuppression therapy (MMF, CTX, CysA, MTX ect) for more than 1 week within 1 month prior to first randomization or intravenous MP Pulse treatment

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Remission rate (complete or partial remission) at 6 months | 6 months after therapy

SECONDARY OUTCOMES:
relapse rate | every 3 months up to 6 months
side effects | every 3 months up to 6 months
  infections, transient increases in serum creatinine, gastrointestinal complaints, liver function disorder and glucose intolerance , etc

CONTACTS AND LOCATIONS:
Overall Officials: Yu Xueqing, MD, Principal Investigator — Department of Nephrology, 1st Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China